CLINICAL TRIAL: NCT05464446
Title: Examination of Lower Urinary System Symptoms and Related Factors in Children With Duchenne Muscular Dystrophy
Brief Title: Examination of Lower Urinary System Symptoms With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Demet Öztürk, Research Assistant, Lokman Hekim University
Other Study IDs: 16969557-1784
Record Dates: First submitted 2022-06-25; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Duchenne Muscular Dystrophy; Lower Urinary Tract Symptoms; Muscle Weakness; Posture Disorders in Children; Lumbar Lordosis; Pelvic Floor Muscle Weakness; Quality of Life
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Lower Urinary Tract Symptoms; Muscle Weakness; Lordosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duchenne Muscular Dystrophy: Children with Duchenne Muscular Dystrophy (DMD) between the ages of 5 and 18 who were diagnosed with DMD by a specialist physician as a result of gene analysis and/or muscle biopsy and their families were included in the study.
  Interventions: Device: Baseline Bubble Inclinometer, Baseline Digital İnclinometer and Hoggan microFET2 devices

INTERVENTIONS:
Device: Baseline Bubble Inclinometer, Baseline Digital İnclinometer and Hoggan microFET2 devices — Bubble inclinometer was used to measure lumbar lordosis angle, Digital inclinometer was used to measure pelvic inclination angle and Hoggan microFET2 was used for muscle strength measurement.

SUMMARY:
The aim of this study is to examine the prevalence of lower urinary tract symptoms (LUTS) in children with Duchenne Muscular Dystrophy (DMD) and the relationship between functional level, posture, muscle strength, pelvic floor muscle control, participation in activities of daily living, and quality of life that may be associated with these symptoms.

Forty-five children with DMD between the ages of 5-18 (Age: 9.00±3.32 years, Weight: 31,10±12,59 kg, Height: 125,87±18,46 cm) and their families were included in the study. LUTS was assessed with Dysfunctional Voiding And Incontinence Scoring System, functional level with Brooke Upper Extremity Functional Classification and Vignos Scale, posture with the New York Posture Assessment Questionnaire, Baseline Bubble Inclinometer (10602, Fabrication Enterprises Inc. New York, USA) and Baseline Digital Inclinometer (12-1057, Fabrication Enterprises Inc, New York, USA), participation in activities of daily living was assessed with the Barthel Index and quality of life was assessed with the Pediatric Quality of Life Inventory 3.0 Neuromuscular Module. Also, using the Hoggan microFET2 (Hoggan Scientific, LLC, Salt Lake City UT, USA) device, hip flexors, quadriceps femoris muscles, shoulder flexors, elbow extensors, elbow flexors, trunk extensors and flexors were evaluated in terms of muscle strength. Evaluations were made once, and the associated factors were compared in the group with and without LUTS, and the relationship between the factors and the severity of LUTS was examined.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with DMD by a specialist physician as a result of gene analysis and/or muscle biopsy,
* Being between the ages of 5-18,
* Volunteering by parents to participate in the study and reading and signing the informed consent form.

Exclusion Criteria:

* Having a diagnosed neuromuscular disease other than DMD and/or with DMD,
* Having a diagnosed psychiatric and/or metabolic disease,
* Having a diagnosis of autism spectrum disorders,
* Presence of congenital and/or acquired anomalies that may affect communication,
* The family and/or the child has a problem of cooperation in completing the assessments for any reason,
* Using a catheter and/or a diaper all day,
* Having difficulty in understanding and speaking the Turkish language.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Duchenne Muscular Dystrophy is an inherited recessive disease linked to the X chromosome. Therefore, only men get the diagnosis, women only become carriers.
Study Population: It consisted of children aged 5-18 years with a diagnosis of DMD and their families.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Lower urinary system symptoms | 1 hour
  It will be investigated how many of the children with DMD participating in the study will have lower urinary system symptoms.
Lower urinary system dysfunction | 1 hour
  It will be investigated how many of the children with DMD participating in the study will have lower urinary system dysfunction.
Muscle strength and lower urinary system symptoms | 1 hour
  It will be investigated whether there is a relationship between lower urinary tract symptoms and muscle strength in children with DMD.
Functionality and lower urinary system symptoms | 1 hour
  It will be investigated whether there is a relationship between lower urinary tract symptoms and functionality in children with DMD.
Posture and lower urinary system symptoms | 1 hour
  It will be investigated whether there is a relationship between lower urinary tract symptoms and posture in children with DMD.
Pelvic floor muscle control and lower urinary system symptoms | 1 hour
  It will be investigated whether there is a relationship between lower urinary tract symptoms and pelvic floor muscle control in children with DMD.
Activities of daily living and lower urinary system symptoms | 1 hour
  It will be investigated whether there is a relationship between lower urinary tract symptoms and activities of daily living in children with DMD.
Quality of life and lower urinary system symptoms | 1 hour
  It will be investigated whether there is a relationship between lower urinary tract symptoms and quality of life in children with DMD.

SECONDARY OUTCOMES:
Urologist evaluation | 1 hour
  It will investigate whether children with DMD have ever been to a urologist in their life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozturk D, Karaduman AA, Akbayrak T. The relationship between lower urinary system symptoms and the level of independence and quality of life in children with Duchenne muscular dystrophy. Pediatr Nephrol. 2024 Oct;39(10):3005-3012. doi: 10.1007/s00467-024-06419-0. Epub 2024 Jun 1. PMID 38822858